CLINICAL TRIAL: NCT04128709
Title: Measurement of Bladder Pressure With a Novel External Device (Cystomanometer) - Home Use
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Christopher Cooper (Other)
Responsible Party: Sponsor-Investigator, Christopher Cooper, Associate Dean, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 201905843
Record Dates: First submitted 2019-10-14; First posted 2019-10-16 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Urinary Bladder, Neurogenic
Keywords: urodynamics; neurogenic; bladder
MeSH Terms: conditions — Urinary Bladder, Neurogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Neurogenic Bladder Patient (Experimental): Patients with neurogenic bladder
  Interventions: Device: Urodynamics Testing

INTERVENTIONS:
Device: Urodynamics Testing — The non-invasive device connects to the end of urinary catheter that the patient uses for routine daily catheterization. Once urine flows into the device the patient presses a single button in order to obtain a pressure measurement which is recorded and stored in the device along with the time and date. The measurement(s) can later be transmitted wirelessly to a smart phone that contains an app for the device.

SUMMARY:
The investigators have developed a novel pressure monitoring device that hooks to standard urinary catheters that are used by patients with a neurogenic bladder on daily clean intermittent catheterization. The device has already been demonstrated to be accurate compared to the gold standard in clinic urodynamics. This study will assess the patients and care givers ability and experience using the device in a home setting.

DETAILED DESCRIPTION:
For patients with neurogenic bladder, regular monitoring of bladder pressure and capacity is a critical component of maintaining renal and urinary health. This monitoring is currently done by in-office urodynamics testing (UDS). This testing is done intermittently, leaving open the possibility of worsening of bladder function and renal deterioration between testing sessions.

This study utilizes a novel pressure monitoring device which is portable and attaches to the end of a standard urinary catheter. The investigators will be investigating if this device can be used by patients or their caregivers in a home setting.

This study will enroll patients with neurogenic bladder that currently perform clean intermittent catheterization on a daily basis as part of their regular care. The patients will be asked to use the device at least twice a day for two weeks.

ELIGIBILITY:
Inclusion Criteria:

* must have diagnosed neurogenic bladder

Exclusion Criteria:

* None

Ages: 1 Year to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-11-19 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Home use of bladder pressure monitoring device | Two weeks
  Utilization study of novel external device

CONTACTS AND LOCATIONS:
Overall Officials: Christopher S Cooper, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospital and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No